CLINICAL TRIAL: NCT01856465
Title: Role of Intestinal Microbiota in Non-alcoholic Fatty Liver Disease Pre and Post bAriatric Surgery
Brief Title: Intestinal Microbiota and NAFLD Pre and Post Bariatric Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Johane Allard (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Johane Allard, Professor of Medicine, Gastroenterologist, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Other Study IDs: 13-6115-A
Record Dates: First submitted 2013-05-14; First posted 2013-05-17 (Estimated); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Morbid Obesity; Non-alcoholic Fatty Liver Disease
Keywords: Bariatric surgery; NAFLD; Steatohepatitis; Simple Steatosis; Intestinal Microbiota
MeSH Terms: conditions — Obesity, Morbid; Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Liver biopsy and stool samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bariatric surgery of morbid obese: Morbid obese patient who undergo Bariatric surgery with NAFLD (NASH or SS) status

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) includes benign hepatic simple steatosis (SS) and steatohepatitis (NASH), which is characterised by inflammation leading to fibrosis and cirrhosis. NAFLD is the hepatic manifestation of the metabolic syndrome, and the prevalence is 74-98% in morbidly obese individuals undergoing bariatric surgery. Although steatosis improves post bariatric surgery, hepatic inflammation and fibrosis do not consistently improve. Alterations of the human gut flora (intestinal microbiota; IM) may play a role. One mechanism linking IM to obesity, insulin resistance (IR), and NAFLD is through translocation of bacterial lipopolisaccharide (LPS=endotoxin) into the blood stream (=endotoxemia), causing chronic inflammation. Morbidly obese subjects have different IM compared to lean controls, and the IM structure is significantly altered after bariatric surgery, probably due to a combination of anatomic changes, diet, and weight loss. For example, the ratio of Firmicutes/Bacteroidetes may be lower in obese subjects compared to lean controls and lower numbers of Faecalibacterium prausnitzii were reported in some obese subjects before bariatric surgery, which increased 3 months post-surgery. This is of interest since, in animal studies, low abundance of F. prausnitzii, a butyrate producing bacterium, is associated with increased intestinal permeability, endotoxemia, and inflammation. To our knowledge, only two studies are available describing IM in patients pre and post bariatric surgery, and no data have been published on the relationship between IM and NAFLD in these patients.

DETAILED DESCRIPTION:
Study Design: A. Cross-sectional study: Sixty patients with morbid obesity undergoing bariatric surgery diagnosed with NAFLD on liver biopsy (30 SS, 30 NASH). Main hypothesis: The ratio of Firmicutes/Bacteroidetes is higher in stool samples from morbidly obese subjects with NASH compared to SS. Other differences in IM composition exist. Objective: to compare bacterial dynamics using Illumina technology to assess the IM. The relative abundance of the dominant fecal microorganisms (including Firmicutes, Archaea, Bacteroides, Bifidobacteria, Mollicutes, Enterobacteriaceae, Clostridia clusters, F. prausnitzii, Roseburia, and Lactobacilli) will also be assessed by real-time PCR. Sub-hypotheses: In NASH compared to SS, there will be: a) lower fecal butyrate concentration; b) higher endotoxin and other inflammatory markers (TNF-α, IL-6) in plasma. Potential covariates assessed: small intestinal bacterial overgrowth (SIBO), measured by glucose hydrogen breath test (GHBT), which can contribute to endotoxemia and inflammation; IR, diabetes status, lipid profile, plasma vitamin E, liver enzymes, anthropometry, food intake, physical activity and environmental factors.

B. Prospective cohort study: Patients undergoing bariatric surgery with either SS or NASH (up to 60 of them recruited from Part A) will be followed prospectively over 12 months to assess changes in the IM and liver histology. Goal is to have 60 subjects who complete the study with a 2nd liver biopsy. Main Hypothesis: In morbidly obese patients with NAFLD (SS or NASH), changes in IM post bariatric surgery will be associated with changes in liver histology. Specifically, an increased number of F. prausnitzii in feces with be associated with improvement in liver histology while a reduction will be associated with deterioration of liver histology. Objective: To correlate changes in liver histology (NAFLD activity score [NAS], inflammation, fibrosis, steatosis) between 0 and 12 months with changes in F. prausnitzii. Other changes of the fecal IM community structure, fecal short chain fatty acids (including butyrate), plasma endotoxin, inflammatory markers (TNF-α, IL-6) and SIBO will also be assessed, in addition to diet, activity, weight change, improvement of diabetes and plasma vitamin E. Secondary hypotheses: Increased number of F. prausnitzii in feces will be associated with increased fecal butyrate, lower serum endotoxin and lower inflammatory markers (TNF-α, IL-6) in plasma.

Significance: In humans with morbid obesity and NAFLD undergoing bariatric surgery, very little data are available on IM and its metabolic effect and contribution to NAFLD. These studies will add more information regarding the role of IM and its effect on potential mechanisms contributing to NAFLD. It will also provide us with pilot data for future intervention studies assessing the potential use of pre- or probiotics for NAFLD in morbidly obese subjects in the setting of bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* BMI>40 kg/m2 or BMI>35-40 kg/m2 with severe weight loss comorbidities
* Male or female, equal or over 18 years of age
* Alcohol consumption is leass than 20 g/d

Exclusion Criteria:

* No diagnosis of NAFLD
* Having liver disease of other etiology
* Having advance liver disease
* Having abnormal coagulation or other reason contraindicating a Liver Biopsy
* On medication known to precipitate steatohepatitis 6 months prior to entry
* On regular intake of non-steroidal anti-inflammatory drugs, prebiotics, probiotics and antibiotics, ursodeoxycholic or any experimental drug in the 3 months prior to study entry
* Having type-1 diabetes, chronic gastrointestinal diseases, previous gastrointestinal surgery modifying the anatomy (prior to bariatric surgery)
* Smoking
* Pregnancy or Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NAFLD is the hepatic manifestation of the metabolic syndrome, and the prevalence is 74-98% in morbidly obese individuals. The aim of this study is to examine the role of intestinal microbiota (IM) in non-alcoholic fatty liver disease (NAFLD) in morbidly obese patients undergoing Roux-en-Y gastric bypass surgery. Alterations of the human gut flora (intestinal microbiota) will be determined before and after surgery in realtion with the change of liver histology.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2013-06 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Firmicutes/Bacteroides ratio in feces | Baseline, 6, 12 months
  16S rRNA sequencing will be performed on the Ion Torrent platform

SECONDARY OUTCOMES:
Overall microbiota composition, amount of selected groups of microorganisms and concentration of Short Chain Fatty Acid (SCFA) in stool sample | 8 months
  Lower fecal butyrate concentration in NASH vs SS
The amount of endotoxin, TNF-alfa and IL-6 in plasma/serum | 8 months
  Higher plasma endotoxin and pro-inflammatory markers (TNF-alfa and IL-6) in NASH vs SS.
The change in inflammation, fibrosis, steatosis in liver histology | 12 months
  Change in the number of F. prausnitzii in stool between baseline and 12 months related with the change in liver histology
NAFLD activity score | baseline, 12 months
  NAFLD Activity score (Kleiner) on liver histology

CONTACTS AND LOCATIONS:
Overall Officials: Johane Allard, MD. FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Mouzaki M, Comelli EM, Arendt BM, Bonengel J, Fung SK, Fischer SE, McGilvray ID, Allard JP. Intestinal microbiota in patients with nonalcoholic fatty liver disease. Hepatology. 2013 Jul;58(1):120-7. doi: 10.1002/hep.26319. Epub 2013 May 14. PMID 23401313
- [Background] Musso G, Gambino R, Cassader M. Recent insights into hepatic lipid metabolism in non-alcoholic fatty liver disease (NAFLD). Prog Lipid Res. 2009 Jan;48(1):1-26. doi: 10.1016/j.plipres.2008.08.001. Epub 2008 Sep 9. PMID 18824034
- [Background] Bellentani S, Scaglioni F, Marino M, Bedogni G. Epidemiology of non-alcoholic fatty liver disease. Dig Dis. 2010;28(1):155-61. doi: 10.1159/000282080. Epub 2010 May 7. PMID 20460905
- [Background] Mathurin P, Hollebecque A, Arnalsteen L, Buob D, Leteurtre E, Caiazzo R, Pigeyre M, Verkindt H, Dharancy S, Louvet A, Romon M, Pattou F. Prospective study of the long-term effects of bariatric surgery on liver injury in patients without advanced disease. Gastroenterology. 2009 Aug;137(2):532-40. doi: 10.1053/j.gastro.2009.04.052. Epub 2009 May 4. PMID 19409898
- [Background] Yang SQ, Lin HZ, Lane MD, Clemens M, Diehl AM. Obesity increases sensitivity to endotoxin liver injury: implications for the pathogenesis of steatohepatitis. Proc Natl Acad Sci U S A. 1997 Mar 18;94(6):2557-62. doi: 10.1073/pnas.94.6.2557. PMID 9122234
- [Background] da Silva VR, Moreira EA, Wilhelm-Filho D, de Miranda JX, Beninca JP, Vigil SV, Moratelli AM, Garlet TR, de Souza Meirelles MS, Vannucchi H, Frode TS. Proinflammatory and oxidative stress markers in patients submitted to Roux-en-Y gastric bypass after 1 year of follow-up. Eur J Clin Nutr. 2012 Aug;66(8):891-9. doi: 10.1038/ejcn.2012.17. Epub 2012 Feb 22. PMID 22353926
- [Background] Musso G, Gambino R, Cassader M. Emerging molecular targets for the treatment of nonalcoholic fatty liver disease. Annu Rev Med. 2010;61:375-92. doi: 10.1146/annurev.med.60.101107.134820. PMID 20059344
- [Background] Frazier TH, DiBaise JK, McClain CJ. Gut microbiota, intestinal permeability, obesity-induced inflammation, and liver injury. JPEN J Parenter Enteral Nutr. 2011 Sep;35(5 Suppl):14S-20S. doi: 10.1177/0148607111413772. Epub 2011 Aug 1. PMID 21807932
- [Background] Spencer MD, Hamp TJ, Reid RW, Fischer LM, Zeisel SH, Fodor AA. Association between composition of the human gastrointestinal microbiome and development of fatty liver with choline deficiency. Gastroenterology. 2011 Mar;140(3):976-86. doi: 10.1053/j.gastro.2010.11.049. Epub 2010 Dec 1. PMID 21129376
- [Background] Ley RE, Turnbaugh PJ, Klein S, Gordon JI. Microbial ecology: human gut microbes associated with obesity. Nature. 2006 Dec 21;444(7122):1022-3. doi: 10.1038/4441022a. PMID 17183309
- [Background] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Background] Duncan SH, Belenguer A, Holtrop G, Johnstone AM, Flint HJ, Lobley GE. Reduced dietary intake of carbohydrates by obese subjects results in decreased concentrations of butyrate and butyrate-producing bacteria in feces. Appl Environ Microbiol. 2007 Feb;73(4):1073-8. doi: 10.1128/AEM.02340-06. Epub 2006 Dec 22. PMID 17189447